CLINICAL TRIAL: NCT07007117
Title: Phase 1 Trial of PHOX2B Peptide-Centric Chimeric Antigen Receptor Autologous T Cells (PHOX2B PC-CAR T) for Relapsed Neuroblastoma
Brief Title: PHOX2B PC-CAR T Cells for Relapsed Neuroblastoma
Acronym: PHOX2B
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stephan Grupp MD PhD (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Alliance for Cancer Gene Therapy (Other); Children's Cancer Research Fund (Other)
Responsible Party: Sponsor-Investigator, Stephan Grupp MD PhD, Chief, Cell Therapy and Transplant Section Director, Susan S. and Stephen P. Kelly Center for Cancer Immunotherapy Medical Director, Cell and Gene Therapy Lab at Children's Hospital of Philadelphia, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-023155; 25CT012 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Refractory Neuroblastoma; Relapsed Neuroblastoma; High-Risk Neuroblastoma
Keywords: Neuroblastoma; PHOX2B PC-CAR T Cells; Cell Therapy
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): The dose escalation arm will determine the maximum tolerated dose of PHOX2B PC-CAR T cells using a standard 3+3 trial design.
  Interventions: Biological: PHOX2B PC-CAR T Cells
- Dose Expansion (Experimental): If at least one dose from the dose expansion arm is determined to be safe, additional patients will be enrolled to the dose expansion arm to preliminarily evaluate the rate of response to PHOX2B-PC CAR T cells and further characterize the safety profile of PHOX2B-PC CAR T Cells
  Interventions: Biological: PHOX2B PC-CAR T Cells

INTERVENTIONS:
Biological: PHOX2B PC-CAR T Cells — The PHOX2B PC-CAR T cell investigational product is comprised of autologous human T cells that have been genetically modified to express a a PHOX2B-targeting chimeric antigen receptor (CAR) transgene.

SUMMARY:
This is a first in human dose escalation trial to determine the safety of administering PHOX2B PC-CAR T cells in patients with advanced, high-risk neuroblastoma.

DETAILED DESCRIPTION:
Neuroblastoma is a tumor of childhood arising from neural crest-derived cells of the developing sympathetic nervous system. While neuroblastomas in young infants often spontaneously regress, children diagnosed with advanced disease after 18 months of age experience poor overall survival despite intensive therapy.

Neuroblastoma is a heterogenous disease, but approximately 50% of patients have a "high-risk" clinical phenotype defined by well-established clinical signs and molecular biomarkers. Over 50% of patients ultimately relapse and survivors are often burdened with significant long-term therapy related morbidities. There is no known cure for patients with relapsed high-risk neuroblastoma. PHOX2B as a therapeutic target for neuroblastoma Paired like homeobox 2B (PHOX2B) is a homeodomain transcription factor that promotes differentiation of neural crest cell derived sympathetic nervous system precursor cells. The PHOX2B protein is so specifically expressed in neuroblastoma that it is used an immunohistochemical confirmation of diagnosis. While PHOX2B is expressed during fetal development, PHOX2B expression is silenced in the vast majority of normal tissues after birth.

To therapeutically leverage this differential expression, an HLA restricted PHOX2B PC-CAR T cell was developed and showed potent inhibition of the growth of neuroblastoma patient-derived xenografts. This investigation will be a single institution, open-label first in human, dose escalation and expansion study designed to assess the safety, tolerability, and manufacturing feasibility of PHOX2B- PC CAR T Cells.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 1 years of age
2. Patients must demonstrate expression of at least one of the following HLA alleles by HLA genotyping (conducted at CHOP) to be eligible:

   HLA-A*24:02, HLA-A*24:03, HLA-A*24:04, HLA-A*24:07, HLA-A*24:124, HLA-A*24:143, HLA-A*24:17, HLA-A*24:242, HLA-A*24:305, HLA-A*24:314, HLA-A*24:33, HLA-A*24:353, HLA-A*24:41, HLA-A*24:51, HLA-A*24:63, HLA-A*24:87, HLA-A*24:92, HLA-A*23:01, HLA-A*23:17, HLA-A*23:25, HLA-A*23:39,
3. Disease Status A. Patients must have high-risk neuroblastoma according to COG risk classification at the time of study enrollment. Patients who were initially considered low- or intermediate-risk, but then reclassified as high-risk are also eligible.

B. Patients must have a previously histologically confirmed diagnosis of neuroblastoma.

C. Patients must have recurrent/progressive, refractory or persistent neuroblastoma.

D. Patients must have neuroblastoma for which standard curative measures do not exist or are no longer effective. Note: Patients at first relapse are eligible as no known curative therapies exist for relapsed high-risk neuroblastoma.

E. Patients must have evaluable or measurable disease at enrollment and at least one of the following:

* Bone Sites

  a) MIBG avid tumors:
  1. Patients with recurrent/progressive or refractory disease:

     a. At least 1 MIBG avid bone site.
  2. Patients with persistent disease:

     1. 3 or more MIBG avid sites (including soft tissue and/or bone).
     2. 1 or 2 MIBG avid sites (including soft tissue and/or bone) with biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one MIBG avid site present at the time of enrollment.

     b) MIBG non-avid tumors: at least 1 bone lesion with either biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma at any time prior to enrollment OR both FDG-PET uptake AND MRI consistent with metastasis.
* Bone marrow: Any amount of tumor cells in the bone marrow (including neuroblasts, mature and maturing ganglion cells).
* Soft tissue site(s) a) At least one soft tissue lesion that meets criteria for a target lesion as defined by: 1. Size: Lesion can be accurately measured in at least one dimension with a longest diameter ≥ 10 mm or for discrete lymph nodes ≥ 15 mm short axis.

  2. In addition to size, a lesion needs to meet ONE of the following criteria:

  a. MIBG avid tumors: i. Patients with recurrent/progressive or refractory disease:

  1. At least one MIBG avid soft tissue site. ii. Patients with persistent disease:
  1. 3 or more MIBG avid sites (including soft tissue and/or bone).
  2. 1 or 2 MIBG avid sites (including soft tissue and/or bone), with biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one MIBG avid site present at the time of enrollment.

     b. MIBG non-avid tumors: biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma (with or without FDG uptake) in a soft tissue site present at time of enrollment OR both FDG-PET uptake AND MRI consistent with metastasis.

     b) At least one soft tissue lesion that does not meet size criteria for a target lesion but had a biopsy positive for neuroblastoma and/or ganglioneuroblastoma at any time prior to enrollment OR is in a patient with recurrent/progressive or refractory disease and is MIBG avid.

  4. Patients must have a Lansky (≤ 16 years) or Karnofsky (> 16 years) score of ≥ 60.

  5. Patients must have adequate renal function defined as age-adjusted serum creatinine ≤1.5 ULN for age.

  6. Liver Function as follows:

  a. Total bilirubin ≤ 1.5 x ULN (exception: total bilirubin ≤ 3 ULN for patients with Gilbert's Disease or liver metastases).

  b. Alanine aminotransferase (ALT) ≤ 3.0 ULN (exception: ALT ≤ 5 x ULN for patients with liver metastases).

  c. Aspartate aminotransferase (AST) ≤ 3.0 ULN (exception: ALT ≤ 5 x ULN for patients with liver metastases).

  7. Pulmonary Function as follows:

  a. Patients need to have a baseline pulse oximetry of at least 92% on room air and DLCO ≥ 60% (corrected for anemia if necessary) if PFTs are clinically appropriate as determined by the treating investigator.

  8. Cardiac Function as follows:

  a. Left ventricular shortening fraction (LVSF) ≥28% or ejection fraction (LVEF) ≥ 50% confirmed by Echo, or adequate ventricular function documented by a scan or a cardiologist.

  9. Patients of child-bearing potential ( patients who have reached menarche and have not experienced treatment-related premature ovarian failure) must have a negative serum pregnancy test performed at the time of screening It is recommended that all patients of reproductive potential use at least one medically acceptable form of contraception for at least 1 year after their last infusion of PHOX2B PC-CAR T cells. Investigators shall counsel patients on the importance of pregnancy prevention and the implications of an unexpected pregnancy.

Exclusion Criteria:

1. Patients with active hepatitis B or active hepatitis C.
2. Patients with active HIV infection (patients undergoing anti-retroviral therapy with undetectable HIV viral load are eligible).
3. Patients with uncontrolled active infection.
4. Patients with primary or acquired immunodeficiency disorder.
5. Concurrent use of systemic steroids or immunosuppression at the time of cell infusion or cell collection, or a condition, in the treating physician's opinion, that is likely to require steroid therapy or immunosuppression during collection or after infusion. Steroids for disease treatment at times other than cell collection or at the time of infusion are permitted. Use of physiologic replacement hydrocortisone or inhaled steroids is permitted as well.
6. Patients with actively progressing CNS metastases, including parenchymal or leptomeningeal involvement. (Note: CNS imaging at screening is only required if there is a clinical indication of suspected CNS metastasis)
7. Active medical disorder that, in the opinion of the investigator, would substantially increase the risk of uncontrollable CRS and/or neurotoxicity.
8. Patients who have received any live vaccines within 30 days prior to enrollment.
9. Pregnant or nursing (lactating) patients.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2032-06-30 (Estimated); Study Completion 2035-06-30 (Estimated)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dose of PHOX2B PC-CAR T Cells | 5 years
  The Maximum Tolerated Dose of PHOX2B-PC CAR T cells will be determined by measuring the incidence of dose limiting toxicities following administration of the product.
Frequency of Adverse Events Following PHOX2B PC-CAR T cell administration | 5 years
  Assess the frequency and severity of treatment related adverse events following administration of PHOX2B PC-CAR T cells.

SECONDARY OUTCOMES:
Manufacturing Feasibility of PHOX2B PC-CAR T cells | 5 years
  Manufacturing Feasibility will be evaluated as the Percentage of patients with PHOX2B PC- CAR T cell products that meet release criteria
Persistence of PHOX2B PC-CAR T cells | 5 years
  Persistence of PHOX2B PC-CAR T cells will be measured by Polymerase Chain Reaction (or flow cytometry) analysis of whole blood to detect and quantify survival of PHOX2B PC-CAR T cells over time.
Preliminarily define the clinical activity of PHOX2B PC-CAR T cells in patients with relapsed or refractory neuroblastoma | 5 years
  Overall Response Rate will be determined based on international Neuroblastoma Response Criteria
Severity of Adverse Events Following Repeated dosing of PHOX2B PC-CAR T Cells | 5 years
  The safety of PHOX2B PC-CAR T cell therapy reinfusions will be measured by the monitoring the frequency and severity of adverse events after multiple PHOX2B PC-CAR T cells infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn Crane, MD, Study Director — Children's Hospital of Philadelphia; Stephan A. Grupp, MD, PhD, Study Director — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States